CLINICAL TRIAL: NCT06040749
Title: Peer-facilitated Virtual Sport for Adults ≥ 50 Years With Spinal Cord Injury
Brief Title: Virtual Sport for Adults ≥ 50 Years With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Kristin Musselman, Principal Investigator, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-5096
Record Dates: First submitted 2023-05-29; First posted 2023-09-18 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-11

CONDITIONS: Spinal Cord Injury
Keywords: Virtual sport; Sport
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual group-based handcycling (Experimental): Virtual group-based handcycling, twice per week for 12 weeks. Each 60-minute session of the intervention will begin with maximum 15 minutes of physiotherapist-led warm-up exercises. Next, a peer-facilitated handcycling session, lasting maximum 45 minutes, will proceed. The handcycling component involves the upper extremities cycling in tandem on a stationary exercise bike. The peer facilitator will be an individual with SCI aged >50 years, who will co-lead participants alongside the physiotherapist through brief group discussion, maximum 40 minutes of moderate-vigorous handcycling, and maximum 5 minutes of cool-down.
  Interventions: Other: Virtual group-based handcycling

INTERVENTIONS:
Other: Virtual group-based handcycling — Virtual group-based handcycling

SUMMARY:
Sport is a physical activity that has many physical, psychological and social benefits for those with spinal cord injury (SCI). However, most sport research involves people with SCI who are <50 years old. This is a problem because many people are >50 years old when first injured. Moreover, people with a SCI are now living longer lives, meaning they also experience more health challenges. Unfortunately, there is limited research studying the impact of sport for adults with SCI aged ≥50 years old.

DETAILED DESCRIPTION:
Aim: To investigate the impact of sport for people with SCI who are ≥50 years old.

Sport Program: This program will be a trial of virtual handcycling. Fifteen male and five female volunteers who are ≥50 years old, ≥12 months post-SCI, wheelchair users, and medically cleared to exercise will be recruited. Five participants will complete the program at a time, as a group, on Microsoft Teams. The sport program will begin with a physiotherapist virtually leading 15 minutes of warm-up exercises. Next, a person living with SCI who is aged ≥50 years old will facilitate 45 minutes of virtual handcycling while screen sharing an indoor cycling application called Zwift, which will provide participants with visual cues and context for changes in exercise intensity. Participants will be provided a cycle ergometer so they can participate in their own homes, and with a smart watch so heart rate can be monitored. This program will run twice a week for three months.

Outcomes: Data will be collected on physical, psychological, and social health at (1) the start of the sport program, (2) immediately after, and (3) three months after the program ends. Any adverse events experienced will be recorded on a survey. Participants' feedback on the sport program and confidence in staying active will also be assessed using an interview at the end.

Conclusion: The knowledge gained will assist in creating future sport programs that may help address the challenges associated with aging and SCI.

ELIGIBILITY:
Inclusion Criteria:

1. Sustained a traumatic or non-progressive, non-traumatic SCI,
2. Chronic stage of recovery (i.e., ≥12 months post-SCI),
3. ≥50 years old,
4. Be a manual wheelchair user,
5. Able to understand spoken English,
6. Can attend two virtual handcycling sessions/week for 12 weeks and attend on-site assessments,
7. Does not intend to change usual physical activity routine throughout duration of the intervention,
8. Be cleared to participate in exercise (determined through completion of the 2022 Physical Activity Readiness Questionnaire for Everyone (PAR-Q+)58),
9. Able to secure hands on handlebars with or without assistance during at-home sessions,
10. Has one emergency contact who can be promptly reached at any point during the intervention,
11. Can independently perform easy-moderate revolutions of arm ergometry movement for ≥10 minutes, with or without adaptations to secure the hands on the handlebars, and
12. Can independently bring up at least one hand to wave at shoulder level.

Exclusion Criteria:

1. Present with significant shoulder pain that reduces use of upper limbs,
2. Present with condition(s) other than SCI that affect ability to use upper limbs or follow English instructions,
3. Have a pressure injury (>grade 2) on the pelvis, sacrum, or hand(s), or
4. Experienced major trauma or surgery within the last 6 months
5. Have a history of cardiovascular disease (myocardial infarction, stroke, hyperlipidemia or untreated hypertension) and do not receive physician clearance to participate.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Spinal Cord Independence Measure | Change from baseline to immediately after the intervention to a 12-week follow-up after the intervention
  A questionnaire that evaluates the functional abilities of individuals with spinal cord injury (SCI). This scale consists of three sub-scales that assess areas of function most relevant to SCI: self-care (scored from 0-20), respiration and sphincter management (scored from 0-40), and mobility (scored from 0-40). Final scores for the Spinal Cord Independence Measure (SCIM) range from 0-100, where a higher score indicates greater functional ability.
Positive Affect and Well-Being Scale of the Quality of Life in Neurological Disorders Measure (PAWB-Neuro-QoL) | Change from baseline to immediately after the intervention to a 12-week follow-up after the intervention
  A questionnaire that assesses affect and sense of well-being. Each statement is to be rated from 1 to 5 ("never" to "always"). The minimum score is 9 and the maximum score is 45. A higher score reflects a greater sense of well-being.
Multidimensional Scale of Perceived Social Support | Change from baseline to immediately after the intervention to a 12-week follow-up after the intervention
  A questionnaire that evaluates perceived help from a significant other, family, and friends. Each statement is to be rated from 1 to 7 ("very strongly disagree" to "very strongly agree"). The minimum score is 12 and the maximum score is 84. A higher score reflects greater perceived social support.
Moorong Self-Efficacy Scale | Change from baseline to immediately after the intervention to a 12-week follow-up after the intervention
  A questionnaire that assesses confidence in performing everyday activities. Each item is scored on a 7-point scale, for a total score out of 112, with a higher score indicating greater self-efficacy.
Spinal Cord Injury Exercise Self-Efficacy Scale | Change from baseline to immediately after the intervention to a 12-week follow-up after the intervention
  A questionnaire that assesses an individual's confidence in performing various physical activities and exercise. Each statement is scored on a 4-point Likert scale, for a total score out of 40, in which a higher score indicates greater perceived exercise self-efficacy.
6 Minute Push Test | Change from baseline to immediately after the intervention to a 12-week follow-up after the intervention
  A field-based assessment that assesses aerobic fitness in manual wheelchair users. During this test, participants will be instructed to propel their wheelchair for 6 minutes along a 30 meter loop while an assessor records the total distanced travelled.
Semi-structured Interview | Within 12 weeks after the intervention
  This interview will explore participants' perspectives on a) whether the intervention affected their physical, psychological, and social health, and b) the delivery of the intervention itself (e.g., components, frequency, duration). A semi-structured interview guide informed by the Modified Health through Sport Conceptual Model will be used as a guide.

SECONDARY OUTCOMES:
Adverse Events | During the 12-week intervention
  Adverse events will be monitored throughout the 12-week intervention. Participants will be asked to complete a survey either online or on paper within 24 hours of experiencing an adverse event. The survey will consist of questions including type, location, and severity. The survey will consist of both closed- and open-ended questions about the circumstances surrounding the adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin E Musselman, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- KITE-Toronto Rehabilitation Institute, UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided